CLINICAL TRIAL: NCT02995447
Title: Differential Effects of Propofol on Scalp and Intracranial Electroencephalogram
Brief Title: Differential Effects of Propofol on Scalp and Intracranial EEG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Martin Soehle, Consultant, University Hospital, Bonn
Other Study IDs: EPI_12
Record Dates: First submitted 2014-10-03; First posted 2016-12-16 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: General Anesthesia
Keywords: propofol; electroencephalogram

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- epilepsy patients: The group consists of patients with therapy refractory epilepsy, in which intracerebral electrodes were implanted to locate the seizure origin and to determine whether the patients are eligible for epilepsy surgery. In an observational study, differences between surface and intracerebral EEG are recorded.
  Interventions: Other: differences between surface and intracerebral EEG

INTERVENTIONS:
Other: differences between surface and intracerebral EEG — No intervention is performed. Im- and explantation of intracerebral electrodes is performed for clinical and not for study purposes. The only difference between study and non-study patients is that the surface as well as the intracerebral EEG is recorded and stored in the former, while it is discarded in the latter.

SUMMARY:
The anesthetic propofol has a dose-depending effect on the EEG, which differs in comparison between scalp and intracerebral electrodes

DETAILED DESCRIPTION:
The electrical activity of the brain (electroencephalogram EEG) is usually assessed from the surface of the head, which is approximately 1-2 cm above the cerebral cortex. Thus, the spatial resolution of the EEG is low, and the electrical activity recorded originates from a multitude of neurons.

Deep brain structures such as the hippocampus also generate electrical activity which cannot be assessed from the surface of the head. However, in some patients electrodes are implanted into the brain to look for the origin of epileptic seizures. Along the way, these intracerebral electrodes enable to record the EEG from intracerebral structures which are generated from few neurons only. Once the origin of epilepsy has been identified, the intracerebral electrodes are removed under general anesthesia.

Anesthetics such as propofol characteristically modify the EEG in a dose-dependant manner. More over, the propofol effect on the EEG recorded from the surface is likely to be different from the intracerebral EEG, however little is known so far. Therefore we aim to investigate the differential effect of propofol on the superficial versus intracerebral recorded EEG.

ELIGIBILITY:
Inclusion Criteria:

* Patients with implanted intracerebral EEG electrodes

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from epilepsy
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2012-11; Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
EEG amplitude | up to two hours of EEG recording
  EEG amplitude in comparison between scalp and intracranial recordings
EEG frequency spectrum | up to two hours of EEG recording
  EEG frequency spectrum in comparison between scalp and intracranial recordings

SECONDARY OUTCOMES:
EEG Burst Suppression Ratio | up to two hours of EEG recording
  EEG Burst Suppression Ratio in comparison between scalp and intracranial recordings

CONTACTS AND LOCATIONS:
Overall Officials: Martin Soehle, MD, PhD, Principal Investigator — Dept. of Anesthesiology and Intensive Care Medicine
Locations (1):
- Dept. of Anaesthesiology and Intensive Care Medicine, University of Bonn, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No